CLINICAL TRIAL: NCT06873880
Title: Integrating Bioelectrical Impedance Analysis and Estimated Glomerular Filtration Rate: A Novel Approach to Assessment of Nutritional Status of Hemodialysis Patients
Brief Title: Integrating BIA and eGFR for Nutritional Status in Hemodialysis Patients
Status: Recruiting | Type: Observational
Sponsor: University of Tartu (Other)
Responsible Party: Principal Investigator, Alastair Forbes, Professor of Medicine, University of Tartu
Other Study IDs: 397/T-10
Record Dates: First submitted 2025-03-04; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: Dialysis; Bioelectrical impedance; Nutrition; Body composition; Renal impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing hemodialysis at Tartu University Hospital: Bioelectrical impedance analysis Background data and clinical findings related to need for dialysis

SUMMARY:
This study looks at how measurements of body composition from Bioelectrical Impedance Analysis (BIA) and estimates of kidney function (eGFR) can be applied together to better assess the health of people on hemodialysis. Many dialysis patients struggle with malnutrition, muscle loss, and fluid imbalances, but current assessment methods rely on unsophisticated tests and observations. By combining BIA and eGFR, this study aims to provide a more accurate and non-invasive way to monitor nutrition and overall health, which could lead to better treatment decisions and improved patient outcomes.

DETAILED DESCRIPTION:
The primary objective of the study is to assess the correlation between Bioelectrical Impedance Analysis (BIA) derived body composition parameters (e.g.fat mass, fat-free mass, total body water, phase angle) and estimated glomerular filtration rate (eGFR) in hemodialysis patients.

The study will investigate how BIA and eGFR can be used together to more effectively monitor nutritional interventions in hemodialysis patients. The study will also assess the prevalence of malnutrition and protein-energy wasting (PEW) in the study population using BIA and eGFR data.

Hemodialysis patients often suffer from complex nutritional problems due to the interplay between renal function, protein-energy wasting and fluid management. Current nutritional assessments in hemodialysis patients are limited, most of which rely on clinical observations or quite basic biochemical tests. A more comprehensive, non-invasive approach is needed to assess both nutritional status and fluid balance. The study will determine whether comparing BIA metrics with eGFR provides a better picture of a patient's nutritional and renal health, which could then improve patient outcomes and dialysis management.

Malnutrition, fluid imbalances, and protein-energy wasting (PEW) are common in patients undergoing hemodialysis due to chronic kidney disease (CKD) and the effects of dialysis therapy. Nutritional status is a critical factor influencing patient outcomes in CKD, but is often under-monitored.

Traditional methods of assessing renal function, such as estimated glomerular filtration rate (eGFR), provide insight into renal health but do not directly measure body composition or nutritional status. Bioelectrical Impedance Analysis (BIA), in contrast, provides a detailed picture of body composition, including fat mass, fat-free mass, total body water, and phase angle. The aim of this study is to investigate the relationship between BIA-derived markers of nutritional status and eGFR to assess their combined utility in assessing nutritional status in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

Chronic kidney disease Hemodialysis for at least 6 months

Exclusion Criteria:

Pregnancy Lactation Major second pathology Pacemaker Recent surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on chronic hemodialysis for at least 6 months
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between body composition and estimated glomerular filtration rate | 3 months
  The primary outcome measure of this study is the correlation between body composition as fat free mass (kg) derived from Bioelectrical Impedance Analysis (BIA) and estimated glomerular filtration rate (eGFR) (ml/minute) in hemodialysis patients.

SECONDARY OUTCOMES:
Assessment of malnutrition in patients on chronic hemodialysis | 3 months
  The study assesses the prevalence of malnutrition and protein-energy wasting (PEW) in the study population using fat-free mass (kg) from BIA and eGFR (ml/minute) data.
Assessment of body composition in patients on chronic hemodialysis | 3 months
  Total body water (ml) derived from BIA will also be compared to the eGFR assessments
Assessment of phase angle in patients on chronic hemodialysis | 3 months
  Phase angle (from BIA) will be compared to the eGFR assessments

CONTACTS AND LOCATIONS:
Overall Officials: Alastair Forbes, MD, Study Director — University of Tartu
Locations (1):
- Institute of Clinical Medicine, Tartu, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: Undecided
Pilot study

REFERENCES:
- [Background] Wang K, Zelnick LR, Chertow GM, Himmelfarb J, Bansal N. Body Composition Changes Following Dialysis Initiation and Cardiovascular and Mortality Outcomes in CRIC (Chronic Renal Insufficiency Cohort): A Bioimpedance Analysis Substudy. Kidney Med. 2021 Feb 18;3(3):327-334.e1. doi: 10.1016/j.xkme.2020.12.008. eCollection 2021 May-Jun. PMID 34136778
- [Background] Bellafronte NT, Vega-Piris L, Cuadrado GB, Chiarello PG. Performance of Bioelectrical Impedance and Anthropometric Predictive Equations for Estimation of Muscle Mass in Chronic Kidney Disease Patients. Front Nutr. 2021 May 21;8:683393. doi: 10.3389/fnut.2021.683393. eCollection 2021. PMID 34095195
- [Background] Guo Y, Zhang M, Ye T, Wang Z, Yao Y. Application of Bioelectrical Impedance Analysis in Nutritional Management of Patients with Chronic Kidney Disease. Nutrients. 2023 Sep 12;15(18):3941. doi: 10.3390/nu15183941. PMID 37764725
- [Background] Son WC, Kwon JG, Hong JP, Park CS, Kim SA, Do JH, Cheon H, Gelvosa MN, Suh HS, Jeon JY. Clinical Utility of Bioelectrical Impedance Analysis Parameters for Evaluating Patients with Lower Limb Lymphedema after Lymphovenous Anastomosis. J Reconstr Microsurg. 2023 Mar;39(3):171-178. doi: 10.1055/s-0042-1750126. Epub 2022 Jul 11. PMID 35817050
- [Background] La Porta E, Faragli A, Herrmann A, Lo Muzio FP, Estienne L, Nigra SG, Bellasi A, Deferrari G, Ricevuti G, Di Somma S, Alogna A. Bioimpedance Analysis in CKD and HF Patients: A Critical Review of Benefits, Limitations, and Future Directions. J Clin Med. 2024 Oct 30;13(21):6502. doi: 10.3390/jcm13216502. PMID 39518641

DOCUMENTS (1):
  • Study Protocol (2025-01-08): https://cdn.clinicaltrials.gov/large-docs/80/NCT06873880/Prot_000.pdf